CLINICAL TRIAL: NCT04843319
Title: Open-Label, Proof-of-Concept and Dose Finding Phase 1b/2 Study of VERU-100 in Men With Advanced Prostate Cancer
Brief Title: To Determine an Effective Dose of VERU-100 for the Treatment of Advanced Prostate Cancer
Acronym: VERU-100
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated as end points were not achieved at current dose level.
Sponsor: Veru Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V2010001
Record Dates: First submitted 2021-04-09; First posted 2021-04-13 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Advanced Prostate Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: Open label single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VERU-100 at various doses (Experimental): 2 ml, 2.5 ml, 3 ml, 3.5 ml of VERU-100
  Interventions: Drug: VERU-100

INTERVENTIONS:
Drug: VERU-100 — GnRH antagonist

SUMMARY:
To determine an effective dose of VERU-100 for the treatment of advanced prostate cancer by assessing its effect on testosterone levels by Day 28 and maintenance through Day 91.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, open-label, dose finding study of VERU-100 to attain and maintain serum total testosterone levels within castrate range (<50ng/dL) in men with advanced prostate cancer. Stage 1 of the study will assess the effect of VERU-100 at various doses. Stage 2 will further assess the efficacy of the effective doses of VERU-100 in an expanded patient population.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years of age
* Be able to communicate effectively with the study personnel
* Have histologically confirmed prostate cancer
* Have prostate cancer staged T3-4NxMx or TxN1Mx or TxNxM1 according to the TNM classification or the patient should have rising PSA after failed local therapy and be candidate for androgen deprivation therapy
* Have a QTc interval <440 ms
* Subjects are judged by the attending physician and/or Principal Investigator to be a candidate for androgen deprivation therapy (continuous therapy)
* ECOG performance status of 0 to 2
* Baseline morning serum testosterone levels >150 ng/dL at Screening Visit
* Have a life expectancy of ≥18 months
* Subjects must agree to use acceptable methods of contraception

  1. If their female partners are pregnant or lactating, acceptable methods of contraception from the time of the first administration of study medication until 6months following administration of the last dose of study medication must be used. Acceptable methods are: Condom used with spermicidal foam/gel/film/cream/suppository. If the subject has undergone surgical sterilization (vasectomy with documentation of azoospermia),a condom with spermicidal foam/gel/film/cream/suppository should be used.
  2. If the male subject's partner could become pregnant, use acceptable methods of contraception from the time of the first administration of study medication until 6 months following administration of the last dose of study medication. Acceptable methods of contraception are as follows: Condom with spermicidal foam/gel/cream/suppository [i.e.,barrier method of contraception], surgical sterilization (vasectomy with documentation of azoospermia) and a barrier method {condom used with spermicidal foam/gel/film/cream/suppository}, the female partner uses oral contraceptives (combination estrogen/progesterone pills), injectable progesterone or subdermal implants and a barrier method (condom used with spermicidal foam/gel/film/cream/suppository).
  3. If the female partner has undergone documented tubal ligation (female sterilization), a barrier method (condom used with spermicidal foam/gel/film/cream/suppository) should also be used.
  4. If the female partner has undergone documented placement of an intrauterine device (IUD) or intrauterine system (IUS),a barrier method (condom with spermicidal foam/gel/film/cream/suppository) should also be used.
* Laboratory values within the following ranges: hemoglobin ≥10 gm/dL, total bilirubin

  * 1.5x upper limit of normal (ULN), AST ≤2.5x ULN, ALT ≤2.5x ULN,
  * 1.5 mg/dL, absolute neutrophil count ≥1500 cell/uL and platelets ≥100,000 cells/uL.
* Creatinine clearance ≥60 mL/min based on Cockcroft-Gault equation.
* Subject is willing to comply with the requirements of the protocol through the end of the study

Exclusion Criteria:

* Prior androgen deprivation therapy within 6 months prior to Screening Visit.
* Potentially curable disease receiving ADT for localized disease
* History of bilateral orchiectomy, adrenalectomy, or hypophysectomy
* Received chemotherapy, cryotherapy, or antiandrogen therapy within 8 weeks prior to the Screening visit for the treatment of prostate cancer.
* Known hypersensitivity to cetrorelix or other LHRH antagonists
* History of Torsade de Pointes
* Currently taking QT-prolonging drugs
* Any disease or condition (medical or surgical) which might compromise the hematologic, cardiovascular, endocrine, pulmonary, renal, gastrointestinal, hepatic, or central nervous system; or other conditions that may interfere with the absorption, distribution, metabolism or excretion of study drug, or would place the subject at increased risk
* Use of exogenous testosterone within 6 months of Screening Visit
* Use of 5α-reductase inhibitor within 3 months of Screening Visit
* Use of systemic corticosteroids at a dose >10 mg/day at Screening
* Major surgery within 4 weeks of Screening Visit (including surgery for prostate cancer)
* Uncontrolled symptomatic congestive heart failure (NYHA Class III -IV), unstable angina pectoris, cardiac arrhythmia, or uncontrolled atrial fibrillation
* History of diabetes mellitus Type 1. Uncontrolled diabetes mellitus Type 2 (control with oral hypoglycemic agents are allowed)
* Received an investigational drug within a period of 90days prior to enrollment in the study
* Received the study medication (VERU-100) previously
* Have been previously diagnosed or treated for active cancer(other than prostate cancer or non-melanoma skin cancer) within the previous five years

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 24 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Percent of men with total testosterone at <50 ng/dL by day 28 | Day 28
  Percent of men that reach castrate level (<50 ng/dL) of total testosterone levels by Day 28

SECONDARY OUTCOMES:
Total testosterone below 20ng/dL levels on VERU-100 | Day 28 and Day 91
  Percent of men that reach <20 ng/dL of total testosterone levels by Day 28 that are maintained at <20 ng/dL through Day 91

CONTACTS AND LOCATIONS:
Overall Officials: Bernette, Study Chair — Veru Inc.
Locations (11):
- United States (11):
  - Arizona Urology Specialist, Tucson, Arizona
  - Urology Associates of Southern Arizona, Tucson, Arizona
  - San Bernardino Urological Associates, San Bernardino, California
  - Genesis Research, LLC, San Diego, California
  - Debbie Urology Johnson, Jeffersonville, Indiana
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Clinical Research Solutions, Middleburg Heights, Ohio
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Houston Metro Urology, Houston, Texas
  - Urology San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No